CLINICAL TRIAL: NCT04154527
Title: Bladder Base Displacement During Abdominal and Pelvic Floor Exercises in Postpartum Women Comparing to Nulliparous Women
Brief Title: Bladder Displacement During Abdominal and Pelvic Floor Exercises
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/610
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Postpartum Disorder
Keywords: pelvic floor; abdominal muscles; ultrasonography; postpartum
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postpartum women with no pelvic floor disorders: This group realised a set of 6 abdominal and pelvic floor exercises, with a muscle recruitment of 25% of maximum force.
  Exercise A: Pelvic Floor contraction Exercise B: Pelvic Floor and Deep Abdominal muscles contraction Exercise C: Pelvic Floor, Deep Abdominal muscles contraction, and axial Stretching Exercise D: Pelvic Floor, Deep and Superficial Abdominal muscles contraction Exercise E: Abdominal Crunch Exercise Exercise F: Low pressure Abdominal Exercise The correct muscle contraction execution was controlled by superficial pelvic floor and abdominal electromyography.
  The bladder base and neck displacement was registered by Transabdominal Ultrasound (TAUS) and Transperineal Ultrasound (TPUS) respectively. To image the bladder base and the bladder neck a 3.5 MHz (megahertz) curved linear array ultrasound transducer was used (LOGIQe Ultrasound,General Electric Healthcare, USA) with the ultrasound unit set in B mode.
  Interventions: Other: Pelvic Floor and Abdominal Exercises
- nulliparous women with no pelvic floor disorders: This group realised a set of 6 abdominal and pelvic floor exercises, with a muscle recruitment of 25% of maximum force.
  Exercise A: Pelvic Floor contraction Exercise B: Pelvic Floor and Deep Abdominal muscles contraction Exercise C: Pelvic Floor, Deep Abdominal muscles contraction, and axial Stretching Exercise D: Pelvic Floor, Deep and Superficial Abdominal muscles contraction Exercise E: Abdominal Crunch Exercise Exercise F: Low pressure Abdominal Exercise The correct muscle contraction execution was controlled by superficial pelvic floor and abdominal electromyography.
  The bladder base and neck displacement was registered by Transabdominal Ultrasound (TAUS) and Transperineal Ultrasound (TPUS) respectively. To image the bladder base and the bladder neck a 3.5 MHz (megahertz)curved linear array ultrasound transducer was used (LOGIQe Ultrasound,GE eneral Electric Healthcare, USA) with the ultrasound unit set in B mode.
  Interventions: Other: Pelvic Floor and Abdominal Exercises

INTERVENTIONS:
Other: Pelvic Floor and Abdominal Exercises — two repetitions of each exercise, during exhalation phase

SUMMARY:
This study evaluates the bladder base displacements during abdominal and pelvic floor exercises in postpartum women comparing to nulliparous women

DETAILED DESCRIPTION:
Postpartum women are at increased risk of suffering pelvic floor dysfunctions. However, only a few researches are focused on the exercises physiological effect at the postpartum recovery period.

A prospective observational study was designed to evaluate the protective or the prolapsed effect of abdominal and pelvic floor exercises in postpartum women.

Two groups were established: Group A was composed of primiparous women during postpartum period and group B of nulliparous women. Both groups practiced the same set of 6 abdominal and perineum exercises. The bladder descent was registered by ultrasonography, and the correct execution was controlled in both groups by superficial pelvic floor and abdominal electromyography.

A Graphical User Interface on MATLAB software has been developed for aiding in offline measurement process.

ELIGIBILITY:
Inclusion Criteria:

* women at postpartum period (more than 6 and less than 12 weeks after vaginal birth)
* willingness to participate in the study
* ability to contract Pelvic Floor Muscles correctly
* written consent to participate.

Exclusion Criteria:

* pregnancy
* caesarean birth
* pelvic Floor disorders
* neurological diseases

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: participants were recruited at the midwife consultation from a Primary Care Health center.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Cranial or Caudal bladder base displacement measured in cm during the set of 6 exercises. | between 6 and 12 weeks after birth
  Cranial or Caudal bladder base displacement during pelvic floor and abdominal exercises, comparing the baseline at rest to the position at 25% of muscle recruitment, in each exercise.
Vertical and horizontal bladder neck displacement measured in cm during the set of 6 exercises. | between 6 and 12 weeks after birth
  Vertical and horizontal displacement of the bladder neck during pelvic floor and abdominal exercises, comparing the baseline at rest to the position at 25% of muscle recruitment in each exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Martinez, PHD student, Principal Investigator — University of A Coruña. Faculty of Physiotherapy, Spain
Locations (1):
- University of Castilla-La Mancha, Toledo, Castille-La Mancha, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available within 6 months after study completion
Access Criteria: Data access will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Thompson JA, O'Sullivan PB, Briffa NK, Neumann P. Comparison of transperineal and transabdominal ultrasound in the assessment of voluntary pelvic floor muscle contractions and functional manoeuvres in continent and incontinent women. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Jul;18(7):779-86. doi: 10.1007/s00192-006-0225-4. Epub 2006 Oct 17. PMID 17043739
- [Background] Barton A, Serrao C, Thompson J, Briffa K. Transabdominal ultrasound to assess pelvic floor muscle performance during abdominal curl in exercising women. Int Urogynecol J. 2015 Dec;26(12):1789-95. doi: 10.1007/s00192-015-2791-9. Epub 2015 Jul 28. PMID 26215905